CLINICAL TRIAL: NCT05694793
Title: Trial for Reliability of Urodynamics SysTem
Acronym: TRUST-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Uro (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-0006; 1R44DK131700 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-06

CONDITIONS: Urologic Diseases; Urodynamics
Keywords: Lower Urinary Tract Dysfunction; Urinary Incontinence; Overactive Bladder; Home Monitoring; Urodynamics; Uroflowmetry
MeSH Terms: conditions — Urologic Diseases; Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Glean Urodynamics System (Experimental)
  Interventions: Device: Glean Urodynamics System

INTERVENTIONS:
Device: Glean Urodynamics System — Wireless, catheter-free urodynamics system
  Other Names: GUS
Device: Glean Urodynamics System — Wireless and catheter free urodynamics system

SUMMARY:
The goal of this prospective trial is to assess the safety and reliability of the Glean Urodynamics System (GUS) in adult females with lower urinary tract symptoms. The main question[s] it aims to answer are:

• What is GUS's ability to safely and reliably conduct wireless, catheter-free monitoring of vesical pressure compared to the vesical pressures collected with conventional urodynamics?

Participants will undergo a conventional urodynamics exam, a simultaneous urodynamics exam with GUS, ambulatory urodynamics with GUS, and extended home monitoring with GUS.

Researchers will compare GUS data with that from a conventional urodynamics exam.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient must be ≥ 18 years of age
2. Patient is a candidate for urodynamics per standard of care
3. Patient or patient's legally authorized representative is able to provide informed consent

Exclusion Criteria:

1. Pregnant (as confirmed by urine pregnancy test or medical history) or breastfeeding, pregnant within the past 6 months or intend to become pregnant during the study period
2. Patient has one or more symptoms indicative of a urinary tract infection (UTI) (i.e., fever, costovertebral angle pain or tenderness, suprapubic tenderness, worsening urinary frequency, worsening urgency, and/or dysuria).
3. Patient has history of recurrent UTIs (≥ 3 episodes in previous 12 months).
4. Patient has used antibiotics within the past 7 days from the baseline/screening visit.
5. Patient diagnosed with neurogenic LUTS (which may be associated with one or more of these conditions: normal-pressure hydrocephalus, cerebral palsy, spinal cord injuries, traumatic brain injury, stroke, Parkinson's disease, multiple sclerosis, meningomyelocele, spina bifida, dementia, Guillain-Barre syndrome, and tumors involving the central nervous systems or spine).
6. Patient diagnosed with interstitial cystitis (IC), bladder pain syndrome, painful bladder syndrome or any etiology of chronic pelvic pain syndrome (CPPS).
7. Patient with a urostomy.
8. Patient has an atypical anatomic structural variation or has had a previous surgical intervention that has permanently changed structural anatomy anywhere along their lower urinary tract (urethra, pelvic floor, urethral sphincter, and/or bladder wall).
9. Patient who has from one or more major strictures in the urethra.
10. Patient has a Pelvic Organ Prolapse Quantification (POP-Q) of Grade III or higher (i.e., most distal portion of the prolapse protrudes more than 1 centimeter below the hymen).
11. Patient with a colostomy.
12. Patient with any abnormal or concerning rectal or vaginal conditions such as ongoing anal fissures, rectocele, fistula, active herpes, active yeast infections, or vaginitis.
13. Patient has a known inability to void or is in complete retention.
14. Subjects who, at the principal investigator's determination, would not be appropriate for this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety | From date of enrollment to study exit (up to 43 days)
  Proportion of participants experiencing a qualifying adverse event attributable to the investigational device

SECONDARY OUTCOMES:
Vesical pressure | during the procedure/surgery
  Vesical pressure

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Tri Valley Urology Medical Group, Murrieta, California
  - University of California San Diego, San Diego, California
  - Unio Health Partners, Torrence, California
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frainey BT, Majerus SJA, Derisavifard S, Lewis KC, Williams AR, Balog BM, Butler RS, Goldman HB, Damaser MS. First in Human Subjects Testing of the UroMonitor: A Catheter-free Wireless Ambulatory Bladder Pressure Monitor. J Urol. 2023 Jul;210(1):186-195. doi: 10.1097/JU.0000000000003451. Epub 2023 Jun 9. PMID 37293725